CLINICAL TRIAL: NCT02742922
Title: Multicenter RCT to Evaluate the Clinical and Cost-effectiveness of a Culturally Adapted Therapy (C-MAP) in Patients With a History of Self-harm
Brief Title: Multicenter Study to Evaluate the Clinical and Cost-effectiveness of a Culturally Adapted Therapy (C-MAP)
Acronym: C-MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other); Dow University of Health Sciences (Other); Karachi Medical and Dental College (Other); Services Hospital, Lahore (Other Government); Peshawar Medical College (Other)
Responsible Party: Principal Investigator, Dr. Nusrat Husain, Chief Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PILL-CMAP-001
Record Dates: First submitted 2016-02-19; First posted 2016-04-19 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Self Harm
Keywords: self harm; culturally adapted therapy; problem solving therapy; low and middle income countries
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culturally adapted therapy (C-MAP) (Experimental): Culturally adapted manual assisted (C-MAP) brief problem solving therapy
  Interventions: Behavioral: Culturally adapted therapy (C-MAP)
- Treatment as usual (No Intervention): This arm will receive no intervention only TAٓU.

INTERVENTIONS:
Behavioral: Culturally adapted therapy (C-MAP) — C-MAP is a brief problem focused therapy, comprising of six sessions delivered within three months. C-MAP is a manual assisted intervention based on the principles of CBT .In this intervention there is an evaluation of the self-harm attempt, crisis skills, problem solving and basic cognitive techniques to manage emotions, negative thinking and relapse prevention strategies.
  Other Names: psycho social intervention
  Arms: Culturally adapted therapy (C-MAP)

SUMMARY:
To evaluate the clinical and cost-effectiveness of a culturally adapted therapy (C-MAP) in patients with a history of self-harm

DETAILED DESCRIPTION:
Suicide is a serious global public health issue, ranked amongst the leading causes of death in many countries. Most of these (75%) are in the low and middle income countries (LAMIC) and globally suicide is the second leading cause of death in young people 15-29 years of age. There is no official data on suicide from Pakistan, a conservative South Asian Islamic country with historically low suicide rates. Both suicide and attempted suicide are illegal acts, as well as socially and religiously condemned, however, there is accumulating evidence that suicide rates have been gradually increasing in Pakistan over the last few years.

The culturally adapted psychological intervention C-MAP utilizes problem solving components within a brief intervention that can be widely utilized in clinical practice. Our previous pilot trial in Karachi shows the efficacy of CBT based intervention(C-MAP) in people who had recently self harmed.The findings from this work have highlighted the applicability of such an intervention to health services in Pakistan for patients who present after a self-harm episode

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 years will be considered eligible for the study.
2. Participants will have to be living within the catchment area of the participating practices and hospitals.
3. Not needing inpatient psychiatric treatment.

Exclusion Criteria:

1. Temporary resident unlikely to be available for follow up.
2. Participants with ICD-I0 mental disorder; due to a general medical condition or substance misuse, dementia, delirium, alcohol or drug dependence, schizophrenia, bipolar disorder, learning disability.
3. Unable to engage, participate or respond to the research questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Suicide Attempt Self Injury Interview SASII | up to 12th months
  Repetition rate of self-harm measured by adapted Suicide Attempt Self-Injury Interview (SASII)

SECONDARY OUTCOMES:
Beck Scale for Suicidal ideation (BSI). | Baseline, 3, 6, 9 and 12th months
  This is a 19-item instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviours, and specificity of a patient's thoughts to kill him/herself during the past week.
Beck Hopelessness Scale | Baseline,3rd,6th,9th and 12th months
  This is a 21 items scale measuring symptoms of depression. Higher scores on the scale indicate greater severity of depression
Beck Depression Inventory (BDI) | Baseline,3rd,6th,9th and 12th months
  This is a 21 items scale measuring symptoms of depression. Higher scores on the scale indicate greater severity of depression
EuroQol-5 Dimensions (EQ5-D) | Baseline,3rd,6th,9th and 12th months
  A standardised instrument to measure health status and associated population utility weights. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression).
Coping Resource Inventory (CRI). | Baseline,3rd,6th,9th and 12th months
  To assess the coping resources to manage stress available to an individual.
Client Satisfaction Questionnaire (CSQ). | Baseline,3rd,6th,9th and 12th months
  The participants will rate their satisfaction with treatment by using the CSQ.

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husian, MD, Principal Investigator — University of Manchester
Locations (7):
- Pakistan (7):
  - Bolan Medical Complex, Quetta, Balochistan
  - Khyber Teaching Hospital, Peshawar, KPK
  - Jinah Hospital, Lahore, Punjab Province
  - Services Hospital, Lahore, Punjab Province
  - Rawalpindi General Hospital, Rawalpindi, Punjab Province
  - Civil Hospital, Karachi, Sindh
  - Abbasi Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Husain N, Kiran T, Chaudhry IB, Williams C, Emsley R, Arshad U, Ansari MA, Bassett P, Bee P, Bhatia MR, Chew-Graham C, Husain MO, Irfan M, Khaliq A, Minhas FA, Naeem F, Naqvi H, Nizami AT, Noureen A, Panagioti M, Rasool G, Saeed S, Bukhari SQ, Tofique S, Zadeh ZF, Zafar SN, Chaudhry N. A culturally adapted manual-assisted problem-solving intervention (CMAP) for adults with a history of self-harm: a multi-centre randomised controlled trial. BMC Med. 2023 Jul 31;21(1):282. doi: 10.1186/s12916-023-02983-8. PMID 37525207
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: Pakistan Institute of Learning and Living — http://pill.org.pk